CLINICAL TRIAL: NCT04717934
Title: Main Study: A Randomized, Evaluator-blinded, No-treatment Controlled, Multicenter Study to Evaluate the Effectiveness and Safety of GAL1906 for Correction of Wrinkles in the décolletage Area Sub-study: A Follow-up Sub-study to Assess Interpretation of Mammograms Following Treatment for Correction of Wrinkles in the Décolletage Area in the Investigational Study 43USRV1906
Brief Title: Main Study: A Study to Evaluate the Effectiveness and Safety of GAL1906 for Correction of Wrinkles in the décolletage Area Sub-study: A Follow-up Study to Evaluate the Analysis of Mammograms Following Treatment for Correction of Wrinkles in Décolletage Area in the Investigational Study 43USRV1906
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USRV1906
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Wrinkle
Keywords: Wrinkles in the Décolletage Area

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- GAL1906 (Experimental): Experimental product for correction of wrinkles
  Interventions: Device: GAL1906
- Control (No Intervention): No treatment control
- Sub-Study (No Intervention): FDA requested extension for mammographic information, which was collected retrospectively as performed per standard of care (not performed as a study intervention)

INTERVENTIONS:
Device: GAL1906 — hyaluronic acid dermal filler gel
  Arms: GAL1906

SUMMARY:
Main study: Randomized, evaluator-blinded, no treatment controlled multicenter study to evaluate safety and effectiveness of GAL1906 for the correction of wrinkles in the décolletage area.

Sub-study: To evaluate imaging interpretation of mammograms in subjects who were enrolled and treated in the 43USRV1906 main study. The sub-study will determine if hyaluronic acid injections in the décolletage interfere with diagnosis or interpretation of mammogram results.

ELIGIBILITY:
Inclusion Criteria for Main study:

* Subjects willing to comply with the requirements of the study and providing a signed written informed consent.
* Non-pregnant, non-breastfeeding females, over the age of 21.
* Subjects seeking treatment for the décolletage.

Inclusion Criteria for Sub-study:

* Subject is willing to comply with the requirements of the study and provide a signed written informed consent.
* Subject has received treatment with GAL1906 in the main protocol.

Exclusion Criteria for Main study:

* Known/previous allergy or hypersensitivity to any injectable HA gel or to gram positive bacterial proteins.
* History of allergy or hypersensitivity to lidocaine or other amidetype anesthetics, or topical anesthetics or nerve blocking agents (if such products are intended to be used for that subject).

Exclusion Criteria for Sub-study:

• Subject is pregnant or nursing AND has no mammogram taken post GAL1906 treatment.

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Main study: The percentage of responders on the Galderma Décolletage Scale, as assessed live by the Blinded Evaluator, at Week 12. | 12 weeks after initial injection
  Responder defined as at least one grade improvement from baseline
Sub-study: Incidence of Breast Image Interference, as Determined by Adjudicated Radiologist | Through the study completion, within 3 months of study start (approximately)
  Incidence of breast image interference, as determined by adjudicated radiologist, leading to potential misdiagnosis due to interference of GAL1906, by evaluation of all performed and collected diagnostic methods as well as comparison of post-treatment mammograms to pretreatment mammograms per subject if applicable.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Galderma Research Site, Birmingham, Alabama
  - Galderma Research Site, Scottsdale, Arizona
  - Galderma Research Site, Redondo Beach, California
  - Galderma Research Site, San Diego, California
  - Galderma Research Site, Vista, California
  - Galderma Research Site, Westport, Connecticut
  - Galderma Research Site, Boynton Beach, Florida
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, Alpharetta, Georgia
  - Galderma Research Site, Chicago, Illinois
  - Galderma Research Site, Baltimore, Maryland
  - Galderma Research Site, New York, New York
  - Galderma Research Site, Spring, Texas
  - Galderma Research Site, Mequon, Wisconsin

IPD SHARING:
Plan to Share IPD: No